CLINICAL TRIAL: NCT06562348
Title: ctDNA Guided Palliative Systemic Therapy Compared to Standard Care in Metastatic Cancer - The Randomized ctDNA-RECIST Trial
Brief Title: The ctDNA-RECIST Trial Part One
Acronym: ctDNA-RECIST
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Karen-Lise Garm Spindler (Other)
Collaborators: Vejle Hospital (Other)
Responsible Party: Sponsor-Investigator, Karen-Lise Garm Spindler, Professor, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KFE 2406
Record Dates: First submitted 2024-08-14; First posted 2024-08-20 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Gastrointestinal Neoplasm
Keywords: Circulating Tumor DNA; Liquid Biopsy; Gastrointestinal Neoplasm; Metastatic
MeSH Terms: conditions — Gastrointestinal Neoplasms; Neoplasm Metastasis | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: An open label 1:1 randomized phase II trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A: Standard of care (Active Comparator): Response evaluation using imaging-based RECIST according to standard guidelines.
  Interventions: Other: Standard of care
- ctDNA-RECIST guided therapy approach (Experimental): Response evaluation will be performed using ctDNA-RECIST instead of imaging.
  Interventions: Other: ctDNA-RECIST guided palliative systemic treatment

INTERVENTIONS:
Other: Standard of care — Patients will be offered palliative systemic treatment according to standard of care. Response evaluation will be performed with the imaging-based RECIST according to standard guidelines. Treatment pauses according to institutional guidelines. Blood samples will be analyzed retrospectively to evaluate ctDNA.
  Arms: A: Standard of care
Other: ctDNA-RECIST guided palliative systemic treatment — Patients are offered palliative systemic treatment according to standard of care. Response evaluation will be performed using ctDNA-RECIST.
  ctDNA is measured before start of treatment. If the baseline sample is ctDNA negative the patient is transferred to an observational cohort, and sampling procedures continues as in the standard arm. If the baseline sample is ctDNA positive the patient continues in the ctDNA-RECIST guided arm. Treatment response is evaluated according to ctDNA-RECIST, and further sampling follows a predefined decision schedule.
  Arms: ctDNA-RECIST guided therapy approach

SUMMARY:
A study investigating if analysis of circulating tumor DNA (ctDNA) can guide palliative treatment in patients with gastrointestinal cancer.

DETAILED DESCRIPTION:
Background:

Circulating tumor DNA, (ctDNA) has the potential to better monitor treatment efficacy compared to imaging, possibly sparing the patient for ineffective treatment and their associated toxicity an allowing for an early change of the treatment approach.

Based on multiple dataset we have defined ctDNA-RECIST - the ctDNA response evaluation criteria.

Aim: This phase II randomized trial evaluates the use of ctDNA Response Evaluation Criteria in Solid Tumors (ctDNA-RECIST) versus standard imaging-based RECIST to guide treatment decisions in patients with metastatic gastrointestinal cancers.

Design: Patients are randomized 1:1. Patients in Arm A are offered standard treatment with response evaluation according to the RECIST criteria based on imaging, and treatment pauses according to institutional guidelines.

In Arm B, treatment response is evaluated based on change in ctDNA between the baseline sample and the evaluation and confirmation sample, according to ctDNA-RECIST:

* Progressive disease: An increase of ctDNA above the previous value with no overlap of the two CI's
* Stable disease: A value within CI of the previous value. The category also includes samples with both previous and present value being 0 (undetectable).
* Partial Response: A decrease below the previous value with no overlap of the two CI'S but the lower CI does not overlap 0.
* Complete response: Decreasing value to an undetectable level
* Near complete response: A decrease below the previous value with no overlap of the two CI'S and with the lower CI overlapping 0

Complete and near complete response can be combined and classified as maximal response.

The study is initiated as a feasibility study (part one)and will continue into the expansion trial after interim analysis.(part two)

ELIGIBILITY:
Inclusion Criteria:

* Incurable metastatic gastrointestinal cancer
* Indication for first or second-line systemic treatment
* Measurable disease according to RECIST v.1.1
* CT of chest and abdomen less than 30 days old at time of treatment initiation
* Age at least 18 years
* ECOG performance status 0-2
* Clinically eligible systemic palliative treatment at investigators decision.
* Adequate bone marrow, liver and renal function allowing systemic chemotherapy
* Anticonception for fertile women and for male patients with a fertile partner. Intrauterine device, vasectomy of a female subject's male partner or hormonal contraceptive are acceptable
* Written and verbally informed consent

Exclusion Criteria:

* Incapacity, frailty, disability and comorbidity to a degree that according to the investigator is not compatible with combination chemotherapy
* Other concurrent malignant tumor except non-melanoma skin cancer or carcinoma in situ cervicis uteri
* Pregnant (positive pregnancy test) or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2029-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Compliance with protocol | 3 months
  The fraction of participants in ARM B, who comply with the study procedures during the first 3 months after inclusion.

SECONDARY OUTCOMES:
Number of treatment cycles | 1 year
  Median number of treatment cycles in the two arms during the first 12 month of stuydy participation
Response rate Arm A | 1 year
  Overall best response and response rate per RECIST during first-line treatment
ctDNA response rate Arm B | 1 year
  Overall best response and response rate per ctDNA-RECIST during first-line treatment

CONTACTS AND LOCATIONS:
Overall Officials: Karen-Lise G Spindler, MD, Prof, Principal Investigator — Department of Oncology, Aarhus University Hospital
Locations (2):
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Department pf Oncology, Vejle Hospital, Vejle